CLINICAL TRIAL: NCT04833270
Title: Pragmatic Randomized Controlled Trial of Non-pharmacological Treatment for Lumbar Disc Herniation : A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Principal Investigator, Kyoung Sun Park, Chief, Clinical study center, Jaseng Hospital of Korean Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-01
Record Dates: First submitted 2021-04-04; First posted 2021-04-06 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Lumbar Disc Prolapse With Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KM non-pharmacological treatment group (Experimental): Non-pharmacological treatment including Korean medicine will be implemented to the participants twice a week for total 8 weeks. The specific intervention will be determined according to the physician's choice, and information will be recorded in the case report form.
  Interventions: Other: KM non-pharmacological treatment group
- Pharmacological treatment group (Active Comparator): Pharmacological treatment will be implemented to the participants twice a week for total 8 weeks. The specific intervention will be determined according to the physician's choice, and information will be recorded in the case report form.
  Interventions: Other: Pharmacological treatment group

INTERVENTIONS:
Other: KM non-pharmacological treatment group — This is a pragmatic setting, and specific intervention is not determined prior to the study. Non-pharmacological treatment including Korean medicine, such as acupuncture, electroacupuncture and chuna, etc, will be chosen by professional physician according to the medical condition of each subject.
  Arms: KM non-pharmacological treatment group
Other: Pharmacological treatment group — This is a pragmatic setting, and specific intervention is not determined prior to the study. The pharmacological treatment will be chosen by professional physician according to the medical condition of each subject.
  Arms: Pharmacological treatment group

SUMMARY:
This is a 2-arm parallel pragmatic randomized controlled trial that will compare non-pharmacological treatment with pharmacological therapy for lumbar disc herniation.

DETAILED DESCRIPTION:
Participants who voluntarily signed informed consent form and eligible for the study were randomly assigned in a 1:1 ratio (15:15) for non-pharmacological treatment and pharmacological treatment group. Participants of each group will receive twice a week for total 8 weeks of intervention. This is a pragmatic randomized controlled trial, so physicians will have medical decision making according to each participant's conditions and choose the specific intervention and dosage of pharmacological and non-pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Numeric rating scale (NRS) score of radiating pain 5 or more for recent 3 serial days.
2. Onset time of radiating pain occurred within 12 weeks.
3. Radiologically diagnosed with lumbar disc herniation in lumbar spine magnetic resonance imaging (L-spine MRI)
4. 19-70 years old
5. participants who agreed and signed informed consent form

Exclusion Criteria:

1. Spine metastasis of cancer, acute fracture of spine, or spine dislocation
2. Progressive neurologic deficits or severe neurologic deficits
3. Soft tissue diseases that can induce low back pain(ie. cancer, fibromyalgia, rheumatoid arthritis, gout,etc)
4. Presence of chronic underlying disease which can interfere the efficacy or interpretation (ie. stroke, myocardial infarct, kidney disease, dementia, diabetic neuropathy, epilepsy, etc)
5. Concurrent use of steroids, immunosuppressants, orpsychotropic medications or any other medication that can interrupt the study result
6. Hemorrhagic disease, severe diabetes or taking anticoagulant drug
7. Participants who took NSAIDs or pharmacopuncture within 1 week
8. Pregnant or lactating women
9. Participants who had undergone lumbar surgery within 3 months
10. Participants who had participated in other clinical trial within 1 month, or have plan for participation in other trial during follow up period of this trial
11. Participants who can not write informed consent
12. Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) of radiating pain in lower extremities | week 9
  NRS is a pain scale in which the patient indicates their subjective pain as awhole number from 0 to 10, where 0 indicates 'no pain or discomfort' and10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of radiating pain in lower extremities | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  NRS is a pain scale in which the patient indicates their subjective pain as awhole number from 0 to 10, where 0 indicates 'no pain or discomfort' and10 indicates 'the most severe pain and discomfort imaginable'.
Numeric rating scale (NRS) of low-back pain | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  NRS is a pain scale in which the patient indicates their subjective pain as awhole number from 0 to 10, where 0 indicates 'no pain or discomfort' and10 indicates 'the most severe pain and discomfort imaginable'.
Visual analogue scale (VAS) of leg radiating pain | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  Visual analogue scale of radiating leg pain, minimum 0 to maximum 100,which is a higher score means a worse outcome.
Visual analogue scale (VAS) of low-back pain | week 1, 2, 3, 4, 5, 6, 7, 8, 9, 14, 27
  Visual analogue scale of radiating leg pain, minimum 0 to maximum 100,which is a higher score means a worse outcome.
Oswestry Disability Index (ODI) | week 1, 5, 9, 14, 27
  ODI is a functional disability questionnaire. The possible range of eachitem score is 0 to 5. Total score range is 0 (better outcome) to 100 (worse outcome)
Fear-Avoidance Beliefs Questionnaire (FABQ) | week 1, 9, 14, 27
  FABQ is one of pateint-reported outcome questionnaire which consists of total 16 questions. Through FABQ, the investigator can evaluate fear avoidance responses, especially in physical and occupational activity domain for patients with low-back pain
Patient Global Impression of Change (PGIC) | week 9, 14, 27
  Participants rate the improvement after treatment on a 7-point Likert scale(1, very much improved; 2, much improved; 3, minimally improved; 4, nochange; 5, minimally worse; 6, much worse; or 7, very much worse.)
Short Form-12 Health Survey version 2 (SF-12 v2) | week 1, 5, 9, 14, 27
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
EuroQol-5 Dimension (EQ-5D-5L) | week 1, 5, 9, 14, 27
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Sun Park, KMD,Ph.D, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No